CLINICAL TRIAL: NCT02187796
Title: PREVALENCE of HIV-ASSOCIATED NEUROCOGNITIVE DISORDERS (HAND) in a SCHOOL of MEDICINE HIV/AIDS OUTPATIENT CLINIC
Acronym: HAND
Status: Completed | Type: Observational
Sponsor: East Tennessee State University (Other)
Collaborators: Neuronetrix, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Norman Moore, Director of Research, Department of Psychiatry, East Tennessee State University
Other Study IDs: 0214.24s
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: HIV-ASSOCIATED NEUROCOGNITIVE DISORDER (HAND)
Keywords: HIV; Dementia; HAND; COGNISION System; ERP; event-related potentials
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Normal Cognition: HIV+ individuals with no detectable neurocognitive impairment
- ANI (asymptomatic neurocognitive impairment): HIV+ individuals where impairment involves at least two cognitive domains, and results in neuropsychological testing performance at least 1 Standard Deviation (SD) below the appropriate mean age/education norm for:
  * Information processing speed
  * Sensory/motor skills
  * Short-term and long-term memory
  * Ability to learn new skills and solve problems
  * Attention, concentration, and distractibility
  * Logical and abstract reasoning functions
  * Ability to understand and express language
  * Visual-spatial organization Visual-motor coordination
  * Planning, synthesizing and organizing abilities
- MCD (Mild Cognitive Disorder): HIV+ individuals with cognitive impairment same as ANI but patient or caregivers report that cognitive deficit interferes with mental acuity, work efficiency, home making or social activity
- HAD (HIV-associated dementia): HIV+ individuals where impairment involves at least two cognitive domains and results in neuropsychological testing at least 2 SD below the appropriate mean age/education norm for:
  * Information processing speed
  * Short-term and long-term memory
  * Ability to learn new skills and solve problems
  * Attention, concentration, and distractibility
  * Logical and abstract reasoning functions
  * Ability to understand and express language
  * Visual-spatial organization Visual-motor coordination
  * Planning, synthesizing and organizing abilities Cognitive impairment significantly interferes with work, home life, social activities or ADL's.
- Healthy Controls (HIV-): Our P300 COGNISION apparatus has been used only in subjects over the age of 60, whereas our participants in the HAND study will all be younger than 60. So, we cannot use COGNISION normative data base for comparison. We will add 10 HIV- healthy controls to our planned 40 HIV+ subjects. These HIV- participants will be age- and gender-matched to the HIV- Asymptomatic Neurocognitive Impairment (ANI) patients, and will undergo all the same assessments

SUMMARY:
1. To determine, in the Quillen College of Medicine HIV+ outpatient clinic, the prevalence of

   * NC (normal cognition )
   * ANI (asymptomatic neurocognitive impairment )
   * MCD (mild cognitive disorder )
   * HAD (HIV-associated dementia )
2. To determine whether the following variables affect the three categories of HAND

   * Time since first diagnosis of HIV infection
   * Anti-viral medications used
   * Age
   * Gender

DETAILED DESCRIPTION:
As life expectancy increases, dementia becomes more common, and the need for its correct diagnosis and treatment becomes more urgent. Alzheimer's disease (AD) is the leading cause of dementia, but its diagnosis is by exclusion of all other causes. Successful treatment of HIV/AIDS has resulted in more patients living long enough to develop HIV-Associated Neurocognitive Disorders (HAND), including dementia.

The National Institute of Mental Health, and the National Institute of Neurological Diseases and Stroke, updated standards for diagnosing HAND. The new criteria created an additional category, HIV-associated asymptomatic neurocognitive impairment (ANI), and modified the name and criteria for what was called MCMD (minor cognitive/motor disorder) to mild cognitive disorder (MCD). HIV-associated dementia (HAD) remained unchanged. Their definition of HAND includes: Cognitive impairment must be attributable to HIV and no other etiology (Dementia, Delirium, Depression, CNS neoplasm, CNS infection other than HIV/AIDS. Cerebrovascular disease, Substance abuse). Their criteria state that cognitive impairment should be validated by neuropsychological testing.

The three categories of HAND are:

1. HIV-associated asymptomatic neurocognitive impairment (ANI)

   Impairment involves at least two cognitive domains, and results in neuropsychological testing performance at least 1 Standard Deviation (SD) below the appropriate mean age/education norm for:
   * Information processing speed
   * Sensory/motor skills
   * Short-term and long-term memory
   * Ability to learn new skills and solve problems
   * Attention, concentration, and distractibility
   * Logical and abstract reasoning functions
   * Ability to understand and express language
   * Visual-spatial organization Visual-motor coordination
   * Planning, synthesizing and organizing abilities
2. Mild Cognitive Disorder (MCD) Same as ANI but patient or caregivers report that cognitive deficit interferes with mental acuity, work efficiency, home making or social activity
3. HIV-associated dementia (HAD)

   Impairment involves at least two cognitive domains and results in neuropsychological testing at least 2 SD below the appropriate mean age/education norm for:
   * Information processing speed
   * Short-term and long-term memory
   * Ability to learn new skills and solve problems
   * Attention, concentration, and distractibility
   * Logical and abstract reasoning functions
   * Ability to understand and express language
   * Visual-spatial organization Visual-motor coordination
   * Planning, synthesizing and organizing abilities Cognitive impairment significantly interferes with work, home life, social activities or ADL's.
4. Non-HIV healthy Controls

Our P300 COGNISION apparatus, provided by Neuronetrix, has been used only in subjects over the age of 60, whereas our participants in the HAND study will all be younger than 60. So, we cannot use COGNISION normative data base for comparison. We will add 10 HIV- healthy controls to our planned 40 HIV+ subjects. These HIV- participants will be age- and gender-matched to the HIV- Asymptomatic Neurocognitive Impairment (ANI) patients, and will undergo all the same assessments

Our IRB-approved study of HAND is limited to neuropsychological assessment. The study could be improved by adding a biological marker assessment, which could help validate the HAND categories. Such a marker is the P300 event-related potential (ERP), known to be related to cognitive processes, such as attention and working memory and abnormal in most neurologic and mental disorders. It could also possibly detect vulnerability to later cognitive impairment in those determined to be of normal cognition by neuropsychological testing. For example, Olichney et al (2011) concluded that ERP studies of individuals at risk for AD may reveal neurophysiological changes prior to clinical deficits, which could advance the early detection and diagnosis of "pre-symptomatic AD". Another example of the association of the P300 and cognition was the study of Onofri et al (2003). In this study donepezil resulted in improved cognition, as measured by a significant increase in MMSE scores. This was accompanied by a reduction of P3 latency. Logistic analysis showed that P3 latency predicted the beneficial effect of donepezil.

ELIGIBILITY:
Inclusion Criteria:

* All participants will have been diagnosed as HIV+.
* Health controls with be age (+/- 5 years) and gender matched to the HIV+ participants.

Exclusion Criteria:

* Alzheimer's DIsease
* Vascular Dementia
* Delirium
* Severe Depression
* CNS Neoplasm
* CNS Infection Other Than HIV/AIDS
* Cerebrovascular Disease
* Alcohol Or Drug Intoxication Or Dependence
* Parkinson's
* Thyroid Disease
* Pernicious Anemia
* Subdural Hematoma
* Occult Hydrocephalus
* Huntington's
* Creutzfeldt-Jakob
* Electroconvulsive Therapy
* Seizure Disorder
* Medical/Psychiatric Disease
* Medication Influencing Cognition

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV+ individuals and Healthy controls (HIV-, age and gender matched)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
IntegNeuro | at enrollment
  IntegNeuro is a touch-screen computerized neuropsychological assessment tool which tests the following cognitive domains:
  * Motor Tapping
  * Choice Reaction Time
  * Time Estimation
  * Word Generation
  * Digit Span
  * Memory recall & Recognition
  * Spot the Word
  * Span of Visual Memory
  * Continuous Performance Test
  * Verbal Interference
  * Switching of Attention
  * Maze
  * Go/No-Go
  * Emotion Processing
IADL (Instrumental Activities of Daily Living Scale) | at enrollment
  HAND criteria include normal activities of daily living for NC and ANI, and impairment of these activities in MCD and HAD. The Instrumental Activities of Daily Living Scale will determine whether the cognitive impairment is interfering with work, home life, social activity or other activities of daily living. The maximum IADL score of 8, means no impairment in any of the following 8 activities; telephoning, shopping, preparing food, housekeeping, laundry, travel, medications and finances. A score of 7 or less will indicate impairment.
Medical Outcomes Study HIV (MOS-HIV) Health Survey | at enrollment
  The Medical Outcomes Study HIV (MOS-HIV) Health Survey is a widely used instrument to assess quality of life in HIV-1-infected individuals. Its cognitive functional status subscale measures functional status owing to neuropsychological (NP) impairment.

SECONDARY OUTCOMES:
MMSE (Mini Mental State Exam) | at enrollment
  The mini-mental state examination (MMSE) or Folstein test is a brief 30-point questionnaire test that is used to screen for cognitive impairment.
COGNISION P300 ODD- BALL DEVICE | at enrollment
  The P300 is evoked by an "oddball' sound of high pitch and irregular timing, compared with sound of lower pitch and regular timing. The subject is asked to count oddball and ignore regular sounds. The P300 is a positive waveform, usually at 300 milliseconds after the oddball sensory input. The COGNISION System is an electroencephalographic (EEG) device that records microvolt level voltage potentials from the subject's scalp. It collects electrophysiological responses to external auditory stimuli, such as in the P300 paradigm. It is composed of (1) a Headset Assembly to be placed on the subject's head at the time of the test, (2) a handheld Headset Control Unit (HCU) to operate the device, (3) computer software to order and monitor the test and analyze the test results, (4) standard stereo earphones (for auditory ERPs).

CONTACTS AND LOCATIONS:
Overall Officials: Norman C Moore, MD, Principal Investigator — Psychiatry and Behavioral Sciences, Quillen College of Medicine, East Tennessee State University; Jonathan P Moorman, MD,Ph.D,FACP, Study Chair — Infectious Diseases, Internal Medicine, Quillen College of Medicine, East Tennessee State University
Locations (1):
- Quillen College of Medicine at East Tennessee State University, Johnson City, Tennessee, United States